CLINICAL TRIAL: NCT00393419
Title: Federal Study of Adherence to Medications in the Elderly (FAME)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: American Society of Health-System Pharmacists (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 04-36002
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2006-10-27 (Estimated); Status verified 2006-10

CONDITIONS: Medication Adherence; Hypertension; Hyperlipidemia
Keywords: hypertension; hyperlipidemia; adherence; pharmacist; elderly; medication
MeSH Terms: conditions — Medication Adherence; Hypertension; Hyperlipidemias

INTERVENTIONS:
Behavioral: Comprehensive pharmacy care program

SUMMARY:
The purpose of this study is to determine the effect of a comprehensive pharmacy care program on medication adherence and persistence, blood pressure, and LDL cholesterol.

DETAILED DESCRIPTION:
Poor medication adherence is prevalent, difficult to manage, and diminishes the health benefits of pharmacotherapies. Elderly patients with coronary risk factors frequently require treatment with multiple medications which places them at increased risk for medication nonadherence. Effective strategies to improve adherence in the elderly are lacking, and improved health outcomes in this population have not been demonstrated.

Objective: We tested the efficacy of a comprehensive pharmacy care program including patient education and an adherence aid (medications custom-packaged in blister packs) to improve medication adherence and its associated effects on blood pressure and low density lipoprotein cholesterol.

This is a Multi-phase, prospective observational and randomized controlled trial. We enrolled community-based patients aged ≥ 65 years old taking ≥ 4 chronic medications per day.

Intervention: After a 2-month run-in phase during which baseline medication adherence (via pill counts), blood pressure, and low-density lipoprotein cholesterol were measured, participants entered a 6-month intervention phase during which standardized medication education and regular follow-up by a clinical pharmacist was provided and medications were dispensed in daily, time-specific blister packs. Following the intervention phase, participants were randomized to continued pharmacy care/blister packs versus usual care (return to their original method of medication administration) for an additional 6 months.

Main Outcome Measures: The primary endpoint of the observation phase was the change in the proportion of pills taken compared to baseline; secondary endpoints were the associated changes in low-density lipoprotein cholesterol and blood pressure. The primary endpoint of the randomized trial was the between-group comparison of medication persistence analyzed according to intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older taking 4 or more chronic medications independently living

Exclusion Criteria:

* assisted living or nursing home residents presence of any serious medical condition for which 1-year survival was expected to be unlikely

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200
Dates: Start 2004-06; Study Completion 2006-08

PRIMARY OUTCOMES:
Change in proportion of pills taken compared to baseline (0-2months) at 8months
Between-group comparison of medication persistence at 14months

SECONDARY OUTCOMES:
Change in blood pressure and low-density lipoprotein cholesterol at 8months

CONTACTS AND LOCATIONS:
Overall Officials: Allen J Taylor, MD, Study Director — Walter Reed Army Medical Center; Jeannie K Lee, Pharm.D, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Blackburn DF, Dobson RT, Blackburn JL, Wilson TW. Cardiovascular morbidity associated with nonadherence to statin therapy. Pharmacotherapy. 2005 Aug;25(8):1035-43. doi: 10.1592/phco.2005.25.8.1035. PMID 16207093
- [Background] Abughosh SM, Kogut SJ, Andrade SE, Larrat P, Gurwitz JH. Persistence with lipid-lowering therapy: influence of the type of lipid-lowering agent and drug benefit plan option in elderly patients. J Manag Care Pharm. 2004 Sep-Oct;10(5):404-11. doi: 10.18553/jmcp.2004.10.5.404. PMID 15369423
- [Background] Jackevicius CA, Mamdani M, Tu JV. Adherence with statin therapy in elderly patients with and without acute coronary syndromes. JAMA. 2002 Jul 24-31;288(4):462-7. doi: 10.1001/jama.288.4.462. PMID 12132976
- [Background] Sokol MC, McGuigan KA, Verbrugge RR, Epstein RS. Impact of medication adherence on hospitalization risk and healthcare cost. Med Care. 2005 Jun;43(6):521-30. doi: 10.1097/01.mlr.0000163641.86870.af. PMID 15908846
- [Derived] Lee JK, Grace KA, Taylor AJ. Effect of a pharmacy care program on medication adherence and persistence, blood pressure, and low-density lipoprotein cholesterol: a randomized controlled trial. JAMA. 2006 Dec 6;296(21):2563-71. doi: 10.1001/jama.296.21.joc60162. Epub 2006 Nov 13. PMID 17101639